CLINICAL TRIAL: NCT07400406
Title: Diagnostic Performance of a Novel Ferumoxytol-enhanced Cardiac Magnetic Resonance for the Detection of Calcified Coronary Arteries: A Single-center Clinical Study.
Brief Title: A Novel Ferumoxytol-enhanced Cardiac Magnetic Resonance for the Detection of Calcified Coronary Arteries
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Chunjian Li, Director of Cardiology, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: 028
Record Dates: First submitted 2026-01-25; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Calcification
Keywords: Ferumoxytol; Magnetic Resonance Imaging; Ultrasmall Superparamagnetic Iron Oxide Particles; Coronary Artery Calcification
MeSH Terms: interventions — Magnetic Iron Oxide Nanoparticles; Ferrosoferric Oxide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with calcified lesions: A novel ferumoxytol-enhanced cardiac magnetic resonance imaging and coronary angiography are performed in patients with CCTA proven calcified lesions occupying greater than 50% of the angle of the vascular lumen.
  Interventions: Drug: Superparamagnetic Iron Oxide Nanoparticles

INTERVENTIONS:
Drug: Superparamagnetic Iron Oxide Nanoparticles — Patients will receive a novel ferumoxytol-enhanced cardiac magnetic resonance imaging.
  Other Names: Ferumoxytol

SUMMARY:
This study is a single-center, prospective, controlled, diagnostic study. The study will be consecutive and is expected to enroll 100 patients with CCTA confirmed coronary calcified lesions. The purpose of this study was to compare the accuracy of novel Ferumoxytol-enhanced Cardiac Magnetic Resonance (Fe-CMR) and coronary CT angiography (CCTA) in detecting calcified coronary arteries, using coronary angiography (CAG) and optical coherence imaging (OCT) as gold standards.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, <75 years;
2. Imaging specialists evaluate CCTA images taken within 30 days and report that calcification occupied one or more of the patient's vascular lumen at an angle of >50% (using the coronary artery segmentation method recommended by the American Heart Association, including nine segments of the major branches of the coronary artery);
3. Patient who will undergo coronary angiography;
4. Patient with normal renal function or chronic renal insufficiency (CKD) stage 1-3;
5. Patient who signs the informed consent.

Exclusion Criteria:

1. People who are allergic to iodine contrast media or have a history of allergy to iron or dextran or are allergic themselves;
2. Because of psychological (such as suffering from claustrophobic syndrome) or physical reasons (such as the presence of metal objects in the body) can not receive MRI examination;
3. suffering from terminal diseases (such as malignant tumors) or life expectancy < 1 year;
4. Pregnant or lactating women;
5. People with limited hearing;
6. Patients with grade III-IV heart function;
7. Patients with a history of coronary artery stent implantation or coronary artery bypass;
8. Other iron agents are being used orally or intravenously;
9. Patients with hemosiderosis or hemochromatosis;
10. Patients with acute coronary syndrome;
11. Patients with hyperthyroidism;
12. Any other candidates deemed unsuitable by the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients with CCTA proven calcified lesions occupying greater than 50% of the angle of the vascular lumen at the First Affiliated Hospital of Nanjing Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Degree of vascular stenosis at the site of coronary calcification. | baseline
  Degree of vascular stenosis at the site of coronary calcification(measured by CAG, CCTA, Fe-CMRA): 0-100%.

SECONDARY OUTCOMES:
CT-FFR, Agatston score, and the angle of calcification lesions occupying vascular lumen | baseline
  ①CT-FFR: computed tomography fractional flow reserve.
  ②Agatston score:0 point: No calcification; 1 to 10 points: Minimal plaque burden; 11 to 100 points: Mild plaque burden; 101 to 400 points: Moderate plaque burden; Greater than 400 points: Extensive plaque burden.
  ③the angle of calcification lesions occupying vascular lumen (CCTA)：0°-360°
calcium score of the plaque measured by OCT | baseline
  OCT: calcium score of the plaque (①Calcification angle: the angle of the calcified plaque surrounding the vessel wall, a larger angle indicates more severe calcification. ②Calcification length: the longitudinal extension length of the calcified plaque along the vessel. ③Calcification thickness: the maximum thickness of the calcified plaque).
Fe-CMRA image quality score | baseline
  Fe-CMRA image quality score: the image quality was assessed by a 4-point scale: 1=poor (coronary vessel barely evident or noisy image); 2=moderate (coronary vessel visible but diagnostic confidence low); 3=good (coronary artery adequately visualized and diagnostic quality image); and 4=excellent (coronary artery clearly depicted).

CONTACTS AND LOCATIONS:
Overall Officials: Chunjian Li, Phd、MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No